CLINICAL TRIAL: NCT03812263
Title: Gene Therapy for Leukocyte Adhesion Deficiency-I (LAD-I): A Phase I/II Clinical Trial to Evaluate the Safety and Efficacy of the Infusion of Autologous Hematopoietic Stem Cells Transduced With a Lentiviral Vector Encoding the ITGB2 Gene
Brief Title: A Clinical Trial to Evaluate the Safety and Efficacy of RP-L201 in Subjects With Leukocyte Adhesion Deficiency-I
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Rocket Pharmaceuticals Inc. (Industry)
Collaborators: California Institute for Regenerative Medicine (CIRM) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RP-L201-0318
Record Dates: First submitted 2019-01-18; First posted 2019-01-23 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Leukocyte Adhesion Defect - Type I
Keywords: Leukocyte Adhesion Deficiency- Type I; LAD-I; ITGB2 mutation; CD18 deficiency
MeSH Terms: conditions — Leukocyte adhesion deficiency type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- RP-L201 (Experimental): RP-L201 is a gene therapy product containing autologous genetically modified CD34+ hematopoietic cells transduced with Chim-CD18-WPRE lentiviral vector administered as a single intravenous infusion
  Interventions: Biological: RP-L201

INTERVENTIONS:
Biological: RP-L201 — CD34+ enriched hematopoietic stem cells from subjects with severe LAD-I transduced ex vivo with lentiviral vector carrying the ITGB2 gene, Chim-CD18-WPRE.

SUMMARY:
The primary purpose of the Phase I portion of the study is to assess the therapeutic safety and preliminary efficacy of a hematopoietic cell-based gene therapy consisting of autologous CD34+ enriched cells transduced with the therapeutic lentiviral vector, Chim-CD18-WPRE, RP-L201. The primary objectives of the Phase II portion of the study are evaluation of survival, as determined by the proportion of subjects alive at age 2 (24 months) and at least 1-year post-infusion without allogeneic hematopoietic stem cell transplant (HSCT) and characterization of the safety and toxicity associated with the infusion.

DETAILED DESCRIPTION:
This is a pediatric non-randomized open-label Phase I/II clinical trial. The Phase I portion will include a safety evaluation and preliminary assessment of the efficacy of hematopoietic gene therapy consisting of autologous CD34+ enriched cells transduced with a lentiviral vector carrying the ITGB2 gene in subjects with severe LAD-I. CD34+ cells will be transduced ex vivo with the therapeutic vector followed by cryopreservation. If the number of CD34+ cells that are available for infusion is at least 2x10e6 total CD34+ cells/kg, subjects will undergo myeloablative conditioning with intravenous busulfan. Subjects will then receive infusion of gene-corrected hematopoietic cells approximately 24 hours following the final busulfan dose.

The active agent is a self-inactivating lentiviral vector carrying the therapeutic ITGB2 gene, encoding for the human CD18 receptor (β2 integrin subunit). The therapeutic product is the subject's autologous hematopoietic stem cells that have been transduced with the lentiviral vector.

ELIGIBILITY:
Inclusion Criteria:

* A confirmed diagnosis of severe LAD-I as demonstrated by flow cytometry indicating CD18 expression on <2% neutrophils (polymorphonuclear neutrophils (PMNs)). Subjects in which CD18+ PMNs are >2% will be considered eligible with <2% CD11a or CD11b expressing PMNs and if there is a documented ITGB2 mutation and clinical history consistent with LAD-I (or known family history).
* At least one (1) prior significant bacterial or fungal infection US NCI CTCAE, v5.0, Grade ≥2). This criterion is not required for subjects with documented family history who meet the above inclusion criteria.
* Age ≥3 months.
* Considered to be an appropriate candidate for autologous transplantation of hematopoietic stem cells.
* A competent custodial parent with legal capacity to execute an institutional review board (IRB)/ethics committee (EC)-approved consent form must be available to participate in the consent process. (Informed assent will be sought from capable subjects, in accordance with the directive of the IRB/EC and with local requirements).
* Ability to comply with trial procedures including investigational therapy and follow-up evaluations.

Exclusion Criteria:

* Availability of a medically-eligible human leukocyte antigen (HLA)-identical sibling donor transplant. Subjects may not be included in this trial as an alternative to a clinically-indicated and feasible HLA-matched sibling donor hematopoietic stem cell transplant. If an HLA-identical sibling is identified, but mobilized peripheral blood or bone marrow hematopoietic stem cell collection is not feasible (for example: donor is in utero, is a newborn from whom cord blood was not collected, or is unable to undergo donation procedure because of medical impairments), then inclusion may be permitted per Investigator discretion.
* Hepatic dysfunction as defined by either:

  * Bilirubin >1.5× the upper limit of normal (ULN) or
  * Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >2.5×ULN.
* Renal dysfunction as defined by either Grade 3 or higher abnormalities in serum sodium, potassium, calcium, magnesium or phosphate as defined by NCI CTCAE v5.0, or the requirement for either peritoneal dialysis or hemodialysis.
* Pulmonary dysfunction as defined by either:

  * Need for supplemental oxygen during the prior 2 weeks (in absence of acute infection).
  * Oxygen saturation (by pulse oximetry) <90%.
* Evidence of active metastatic or locoregionally advanced malignancy (including hematologic malignancy) for which survival is anticipated to be less than 3 years.
* Serious infections with persistent bloodstream pathogens at time of trial entry. (Subjects with active infections (e.g., unresolved ulcerative lesions, skin or oral infections) are permitted as long as appropriate antibiotic therapy has been (or is being) administered).
* Any medical or other contraindication for both leukapheresis and bone marrow harvest procedure, as determined by the treating Investigator.
* Any medical or other contraindication for the administration of conditioning therapy, as determined by the treating Investigator.
* Significant medical conditions, including documented human immunodeficiency virus (HIV) infection, poorly-controlled diabetes, poorly-controlled hypertension, poorly-controlled cardiac arrhythmia or congestive heart failure; or arterial thromboembolic events (including stroke or myocardial infarction) within the 6 prior months.
* Any medical or psychiatric condition that in the opinion of the Investigator renders the subject unfit for trial participation or at higher than acceptable risk for participation.

Min Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-08-30 (Actual); Primary Completion 2023-09-12 (Actual); Study Completion 2023-09-12 (Actual)

PRIMARY OUTCOMES:
Phase I: Number of participants with treatment-related adverse events as assessed by United States (US) National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v.5.0 | 2 years
  Evaluation of safety associated with treatment with RP-L201
Phase II: Survival following infusion of RP-L201 | 2 years
  , as determined by the proportion of subjects alive at least 1-year post investigational product infusion without allogeneic HSCT and alive at age 2 (24 months) without allogeneic HSCT for subjects less than 1 year of age at study enrollment.
Phase II: Number of participants with treatment-related adverse events as assessed by CTCAE v.5.0 | 2 years
  Evaluation of safety associated with treatment with RP-L201

SECONDARY OUTCOMES:
CD18 expression after infusion of RP-L201 | 2 years
  Determination of the percentage of subjects in whom infusion of RP-L201 results in a change in the percentage of neutrophils expressing CD18 to at least 10%
Genetic correction after infusion of RP-L201 | 2 years
  Determination of the percentage of subjects in whom infusion of RP-L201 results in at least 10% of peripheral blood neutrophils carrying the therapeutic Chim-CD18-WPRE lentiviral vector provirus at 6 months post-infusion
Incidence of infections after infusion of RP-L201 | 2 years
  Determination of the incidence of significant infections, infection-related hospitalizations, and prolonged infection-related hospitalizations, comparing the incidences prior to investigational product infusion and subsequent to hematopoietic reconstitution.
Assessment of LAD-I-associated neutrophilia after infusion of RP-L201 | 2 years
  Evaluation of change to partially normal or to normal levels of LAD-I-associated neutrophilia
Assessment of LAD-I-associated leukocytosis after infusion of RP-L201 | 2 years
  Evaluation of change to partially normal or to normal levels of LAD-I-associated leukocytosis
Assessment of skin rash or periodontal abnormalities after infusion of RP-L201 | 2 years
  Evaluation of resolution (partial or complete) of any underlying skin rash or periodontal abnormalities
Assessment of overall survival after infusion of RP-L201 | 2 years
  Assessment of event-free survival (EFS) defined as survival without graft failure (GF) and without acute graft-versus-host disease (aGVHD) grade 2 to 4.

CONTACTS AND LOCATIONS:
Overall Officials: Donald B Kohn, MD, Principal Investigator — University of California, Los Angeles; Claire Booth, MBBS, PhD, MSc, Principal Investigator — University College London Great Ormond Street Institute of Child Health; Julián Sevilla Navarro, MD, PhD, Principal Investigator — Hospital Infantil Universitario Niño Jesús
Locations (3):
- University of California, Los Angeles, Los Angeles, California, United States
- Hospital Infantil Universitario Niño Jesús (HIUNJ), Madrid, Spain
- University College London Great Ormond Street Institute of Child Health, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Booth C, Sevilla J, Almarza E, Kuo CY, Zubicaray J, Terrazas D, O'Toole G, Chitty-Lopez M, Choi G, Nicoletti E, Long-Boyle J, Fernandes A, Chetty K, De Oliveira S, Banuelos C, Xu-Bayford J, Bastone AL, John-Neek P, Jackson C, Moore TB, Gilmour K, Schambach A, Rothe M, Kasbekar S, Rao GR, Patel K, Shah G, Thrasher AJ, Bueren JA, Schwartz JD, Kohn DB. Lentiviral Gene Therapy for Severe Leukocyte Adhesion Deficiency Type 1. N Engl J Med. 2025 May 1;392(17):1698-1709. doi: 10.1056/NEJMoa2407376. PMID 40305711